CLINICAL TRIAL: NCT03367026
Title: Reducing Elevated Heart Rate in Patients With Severe Sepsis by by the "Funny Channel" Current (If) Inhibitor Ivabradine
Brief Title: Reducing Elevated Heart Rate in Patients With Severe Sepsis by Ivabradine
Acronym: REHSI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REHSI
Record Dates: First submitted 2017-10-01; First posted 2017-12-08 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-10

CONDITIONS: Sepsis, Severe
Keywords: ivabradine; sepsis; heart rate
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ivabradine oral product (Active Comparator): Patients in the ivabradine treatment arm receive interventions:an additional enteral preparation (orally, via nasogastric tube or Jejunum tube) of ivabradine for 4 days.
  Interventions: Drug: Ivabradine Oral Product
- control group (No Intervention): All patients receive established medical therapy according to current guidelines and therapeutic standards.

INTERVENTIONS:
Drug: Ivabradine Oral Product — Patients in the ivabradine treatment arm receive an additional enteral preparation (orally, via nasogastric tube or Jejunum tube) of ivabradine for 4 days.
  Day 1 :
  2.5 mg ivabradine b.i.d. if heart rate ≥90 bpm
  Day 2,3,4:
  2.5 mg ivabradine b.i.d. if 60bpm≥heart rate<90bpm. 5.0mg ivabradine b.i.d. if heart rate ≥90bpm
  Other Names: routine therapy
  Arms: Ivabradine oral product

SUMMARY:
REHSI is a prospective, multi-center, open label, randomized, controlled two arms, to evaluate the ability of ivabradine to reduce an elevated heart rate in septic shock patients. The primary end point is the reduction of heart rate within 24 hours. This trial will randomize 70 patients (men and women, aged ≥ 18 years) with newly diagnosed Septic Shock (despite adequate fluid resuscitation, were still requiring high-dose norepinephrine (NE) to maintain a mean arterial pressure (MAP) ≥65 mmHg , and had a tachycardia >100 beats per minute (bpm). Treatment period will last 4 days. All patients will be followed for up to six months.

ELIGIBILITY:
Inclusion Criteria:

1. Severe sepsis due to coronary and non-coronary etiology
2. Severe sepsis diagnosed ≤ 24 h
3. Sinus rhythm with heart rate ≥ 100bpm
4. Written informed consent or identified or suspected positive will with respect to the trial treatment

Exclusion Criteria:

1. Patients who have not yet completed the 18th year of age
2. Pregnancy, lactation
3. Patients with a history of pre-existing chronic renal failure with a glomerular filtration rate <30ml/min
4. severe hepatic insufficiency
5. Sick sinus syndrome
6. Sinu-atrial block
7. pacemaker-dependency 8.3rd degree AV block

9.Use of potent cytochrome P450 3A4 inhibitors such as antifungals of the azole -type (ketoconazole, itraconazole), macrolide antibiotics (clarithromycin, erythromycin per os, josamycin, telithromycin), HIV protease inhibitors (nelfinavir, ritonavir) and nefazodone (see Summary of Product Characteristics (SPC))

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
mean heart rate | 24 hours
  the reduction of the mean heart rate of 24 hours after the start of trial treatment

SECONDARY OUTCOMES:
severity of illness | 4 days
  measured by serial APACHE II score monitoring and Sequential Organ Failure Sequential Organ Failure Assessment (SOFA) score monitoringAssessment (SOFA) score monitoring
mean heart rate | 4 days
  comparison of the mean heart rate between the treatment and control group
mortality | 6 months
  28-day and 6 months mortality